CLINICAL TRIAL: NCT06710938
Title: Exploratory Study of Thoracoabdominal Artery Stent Graft System in the Treatment of Thoracoabdominal Aortic Aneurysms
Brief Title: Thoracoabdominal Artery Stent Graft System Exploratory Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: LT/TS-TAAA-EU-01
Record Dates: First submitted 2024-11-15; First posted 2024-11-29 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Thoracoabdominal Aortic Aneurysms
Keywords: Thoracoabdominal Aortic Aneurysms; G-branch Stent Graft; Lifetech Scientific; Thoracoabdominal Artery Stent Graft System
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Intervention Model Description: Thoracoabdominal Artery Stent Graft System. The system includes the G-Branch™ thoracoabdominal aortic stent graft system, the peripheral vascular stent graft system, and the aortic extension stent graft system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endovascular therapy used as treatment of TAAA (Experimental): Traditional methods of treatment of TAAA include open surgery and hybrid surgery. Open surgery requires Thoracoabdominal incision which will result in a huge wound and the reconstruction of the visceral artery is also complicated. endovascular therapy has been developed for many years and has demonstrated significant advantages, such as small wounds, and fewer complications. Now Endovascular therapy is gradually used in the treatment of TAAA as well. Compared with traditional open surgery and hybrid surgery, the risk-benefit ratio of endovascular therapy is much better. When the risk-benefit gap between the investigational device and existing treatments is so wide that a control group is ethically unfeasible. So a single-arm exploratory study is adopted.
  Interventions: Device: The system includes the G-Branch™ thoracoabdominal aortic stent graft system, the peripheral vascular stent graft system, and the aortic extension stent graft system

INTERVENTIONS:
Device: The system includes the G-Branch™ thoracoabdominal aortic stent graft system, the peripheral vascular stent graft system, and the aortic extension stent graft system — The thoracoabdominal artery stent graft system is a mixed branch design with two inner branches for the visceral arteries and two outer branches for the bilateral renal arteries.

SUMMARY:
This study is designed as a single-center, prospective, single-arm, open-label, exploratory study. The objective is to evaluate the feasibility of Thoracoabdominal Artery Stent Graft System for endovascular treatment of Thoracoabdominal aortic aneurysms (TAAA).

DETAILED DESCRIPTION:
Thoracoabdominal Aortic Aneurysms involve both thoracic and abdominal aortic arteries, as well as abdominal aortic aneurysms above the renal arteries. The treatment of TAAAs is complicated because the disease involves multiple visceral arteries. Traditional methods of treatment of TAAA include open surgery and hybrid surgery. The early postoperative mortality, as well as postoperative complications such as respiratory failure, renal failure, and other vital organ complications are concern for open surgery, which makes the benefit-risk ratio of traditional open surgery remains unsatisfactory. In addition, open surgery requires thoracoabdominal incision which will result in huge wound and the reconstruction of visceral artery is also complicated. Hybrid surgery, comprised of an initial open visceral debranching procedure followed by endovascular aneurysm exclusion, is another treatment option. Although hybrid surgery can reduce the huge wound caused by thoracotomy, it does not seem to result in lower complication rates at early and midterm follow up.

With the rapid development of endovascular treatment technology, endovascular therapy is also applied in the treatment of TAAA, and gradually becomes one of the main treatment method. Especially for patients with high surgical risk because of comorbidities, an endovascular solution may be preferable. Total endovascular aneurysm repair (t-EVAR) without debranching surgery does not require thoracotomy and laparotomy and could improve the outcomes of these patients. t-EVAR includes fenestrated EVAR (f-EVAR), multi-branched EVAR (b-EVAR), and physician-modified fenestration endograft (PMFG). Compared with open surgery and hybrid surgery, endovascular therapy has the following advantages: 1) minimally invasive surgery, avoiding thoracic and abdominal incision; 2) avoiding aorta occlusion during the operation so that reduce various visceral ischemia complications; 3) reducing intraoperative blood loss and hospital stay; 4) reducing spinal cord complications.

The TAAA stent graft system used for endovascular treatment generally consists of a stent graft and a delivery system. Stent graft, also known as artificial stent-type vascular graft, is generally composed of tubular covered and metal wire braided stent. The stent can be compressed into the sheath which delivers the stent to the lesion site of TAAA, and then is released from the sheath. The stent opens by its own expansion force to separate the blood from the lesion site, so as to achieve the treatment purpose. Custom made stents need to be designed and manufactured according to the patient's aortic characteristics, and the 6-8 week waiting period limits its use in patients who show precursors to rupture or who have already ruptured. Currently commercially available off-the-shelf multibranched stent grafts for TAAA include Zenith t-Branch stent (Cook), E-nside TAAA Multibranch Stent Graft System (Jotec) and GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis (Gore & Associates). A critical issue with these multibranched stent grafts is the limited device specification and suboptimal anatomical feasibility for TAAA patients, therefore, improvements to the device profile, configuration and size optimization are needed. In the current context, Lifetech have developed a new TAAA stent graft system, Thoracoabdominal Artery Stent Graft System, which is a mixed branch design with two inner branches for the visceral arteries and two outer branches for the bilateral renal arteries. It is an off-the-shelf multibranched endograft and there is no need to waste time on customisation. The variations in the main body diameter, length and branch size, introducing diversified configurations that accommodate more anatomic conditions. Two inner branches are integrated with preloaded guidewires to facilitate visceral artery cannulation and reduce the procedure time. The semi-release design allows the stent position to be adjusted during the release process, making the stent positioning more accurate and less difficult.

This study is an exploratory study aimed to assess the feasibility of the Thoracoabdominal Artery Stent Graft System.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 80 years old;
2. Patients diagnosed with a Thoracoabdominal aortic aneurysm (based on the modified Crawford classification and European Society for Vascular Surgery (ESVS) 2019 Clinical Practice Guidelines on the Management of Abdominal Aorto-iliac Artery Aneurysms), and should meet at least ONE of the following conditions:

   1. Maximum diameter of TAAA is >50 mm;
   2. TAAA diameter increases by more than 5 mm in the past 6 months or by more than 10 mm in the past 1 year;
   3. Definite symptoms associated with TAAA, such as abdominal pain and back pain.
3. Anatomical Criteria

   1. Proximal landing zone (aorta or implanted graft): the diameter ranges from 17 to 36 mm, and length should be ≥25 mm;
   2. Distal landing zone (aorta or implanted graft): If distal landing zone is in iliac artery, distal landing zone diameter ranges from 7 to 25 mm, and length should be ≥15 mm; If the distal landing zone is in the abdominal aorta, distal landing zone diameter ranges from 12 to 36 mm, and length should be ≥20 mm.
   3. Visceral branch landing zone: the diameter ranges from 6 to 13 mm, and the length should be ≥15 mm;
   4. Renal artery landing zone: the diameter ranges from 4.5 to 9 mm, and the length should be ≥15 mm;
   5. Appropriate iliac, femoral, and upper limb arterial access.
4. Patients who understand the purpose of the study, volunteer to participate and sign the informed consent form, and are willing to complete follow-up as required by the protocol;
5. Patients do not want to or cannot wait for the approved alternative

Exclusion Criteria:

Exclusion Criteria (not eligible if any of the criteria is met):

1. Patients with ruptured thoracoabdominal aortic aneurysms in unstable hemodynamic condition;
2. Patients with thoracoabdominal aortic dissection;
3. Patients with infected or mycotic thoracoabdominal aortic aneurysms;
4. Patients with systemic or local infections that may increase the risk of endovascular graft infection;
5. Patients with occluded superior mesenteric artery, celiac trunk artery, or renal artery;
6. Patients requiring simultaneous coverage or embolization of bilateral internal iliac arteries;
7. Patients with severe stenosis, calcification or mural thrombus at stent-graft landing zone, and this situation leads to difficulty in adhering the covered stent or affecting the patency of the stent;
8. Patients with a history of acute coronary syndrome within the recent 6 months; Acute coronary syndrome refers to acute cardiac ischemic syndrome caused by rupture or erosion of unstable atherosclerotic plaques in the coronary artery and fresh thrombosis, including ST-segment elevation myocardial infarction (STEMI), non-ST-segment elevation myocardial infarction (NSTEMI) and unstable angina pectoris.
9. Patients with transient ischemic attack (TIA) or ischemic/hemorrhagic stroke within the recent 3 months;
10. Patients with abnormal liver and kidney function before operation [alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the upper limit of normal value; Serum creatinine (Cr) >150umol/L];
11. Patients with severe pulmonary insufficiency who cannot tolerate general anesthesia;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2031-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Treatment success rate | Intraoperative and 12-month post operation
  Treatment success is a composite index that should meet all of the following criteria:
  * Immediate technical success: refers to successful delivery of the delivery system to the intended location, successful deployment of the stent graft, withdrawal of the delivery system, with no type I/III endoleak) [Timeframe: intraoperative],
  * No TAAA-related secondary intervention (including secondary intervention due to aneurysm rupture, sustained enlargement, stent migration, type I/III endoleak, branch stenosis/occlusion) [Timeframe: 12-month post operation].
Incidence of major adverse events (MAEs): 30-day post operation | 30-day post operation
  MAEs are defined as all-cause death, hepatic failure, bowel necrosis, renal failure, stroke, permanent paraplegia, myocardial infarction, and respiratory failure.

SECONDARY OUTCOMES:
Incidence of perioperative delivery system-related complications | intraoperative and within 30-day post operation
  Include conversion to open surgery, hemorrhage, hematoma, and pseudoaneurysm of the atrial access.
All-cause mortality | 6-month, 12-month, and 2- to 5-year post operation
  All-cause death is defined as death from any cause during the follow-up period.
TAAA-related mortality | 6-month, 12-month, and 2- to 5-year post operation
  TAAA-related death is defined as death due to rupture of TAAA or surgical treatment of TAAA.
Incidence of serious adverse events (SAEs) | 6-month, 12-month, and 2- to 5-year post operation
  If staged reconstruction is performed because of the patient's condition, then the reconstruction should not be a serious adverse event.
Incidence of device-related adverse events | 6-month, 12-month, and 2- to 5-year post operation
  Adverse events refer to adverse medical events that occur during a clinical trial, regardless of whether they are related to the investigational device. However, normal postoperative stress reactions, such as fever and constipation, should be distinguished. If events are judged by the investigator as normal postoperative stress reactions, they need not be recorded as adverse events. If staged reconstruction is chosen because of the patient's condition, then the reconstruction should not be an adverse event.
Incidence of increase in maximum diameter of aneurysm >5mm | 6-month, 12-month post operation
Incidence of type I or III endoleaks | 6-month, 12-month post operation
Incidence of stent graft migration | 6-month, 12-month post operation
  The evaluation criteria are as follows: 1) the stent graft migration at the follow-up point after operation is more than 10mm compared with the position before discharge, or 2) the migration caused symptoms or required intervention.
Patency rate of branch vessels | 6-month, 12-month post operation
  Patency of branch vessels is defined as stenosis ≤50% of the branch vessels.
Incidence of TAAA-related secondary intervention | 6-month, 12-month, and 2- to 5-year post operation
  If staged reconstruction is performed because of the patient's condition, then the reconstruction should not be a secondary intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Asklepios Klinik Nord Heidberg, Hamburg, Germany